CLINICAL TRIAL: NCT01257516
Title: An Open-Label, Multiple-Dose, Randomized, 2-Way Crossover Study In Healthy Volunteers To Determine The Steady-State Pharmacokinetics Of 660 Mg (2 X 330 Mg Tablets) Pregabalin Controlled Release Formulation Administered Following An Evening Meal Relative To The 300 Mg Of The Immediate Release Formulation Administered Twice Daily
Brief Title: An Investigation Of The Absorption And Pharmacokinetics Of Multiple Doses Of A Controlled Release Pregabalin Tablet As Compared To Multiple Doses Of The Immediate Release Pregabalin Capsule In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081216
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-03

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin immediate release, 300 mg (Other): Reference Treatment
  Interventions: Drug: Pregabalin immediate release, 300 mg
- Pregabalin controlled release, 330 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg

INTERVENTIONS:
Drug: Pregabalin immediate release, 300 mg — 300 mg immediate release capsule administered twice daily for four days
  Arms: Pregabalin immediate release, 300 mg
Drug: Pregabalin controlled release, 330 mg — Two tablets of 330 mg (total dose of 660 mg) given concurrently once daily for four days
  Arms: Pregabalin controlled release, 330 mg

SUMMARY:
The purpose of this study is to 1)evaluate the extent of absorption of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of the pregabalin immediate release capsule, 2) evaluate the pharmacokinetics of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of pregabalin immediate release capsule and 3) evaluate the safety and tolerability of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of the pregabalin immediate release capsule.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of pregabalin immediate release capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve at steady-state over a 24 hour period (AUC24)for assessment of equivalence between 330 mg CR (two tablets administered concurrently for a total 660 mg dose) and 300 mg IR capsule given 2times daily (total daily dose 600 mg) | 5 days

SECONDARY OUTCOMES:
Safety endpoints include evaluation of adverse events | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Chew ML, Alvey CW, Plotka A, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pregabalin controlled-release pharmacokinetics in healthy volunteers: analysis of four multiple-dose randomized clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):627-37. doi: 10.1007/s40261-014-0221-2. PMID 25078977
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081216&StudyName=An%20Investigation%20Of%20The%20Absorption%20And%20Pharmacokinetics%20Of%20Multiple%20Doses%20Of%20A%20Controlled%20Release%20Pregabalin%20Tablet%20As%20Compared%20To%20Multi